CLINICAL TRIAL: NCT02431559
Title: Phase 1/2 Study of Chemoimmunotherapy With Toll-like Receptor 8 Agonist Motolimod (VTX-2337) + Anti-PD-L1 Antibody MEDI4736 in Subjects With Recurrent, Platinum-Resistant Ovarian Cancer for Whom Pegylated Liposomal Doxorubicin is Indicated
Brief Title: Phase 1/2 Study of Motolimod, Doxorubicin, and Durvalumab in Recurrent, Platinum-Resistant Ovarian Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ludwig Institute for Cancer Research (Other)
Collaborators: MedImmune LLC (Industry); Celgene (Industry); Cancer Research Institute, New York City (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: LUD2014-001
Record Dates: First submitted 2015-04-27; First posted 2015-05-01 (Estimated); Results first posted 2019-09-23 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-10

CONDITIONS: Ovarian Cancer
Keywords: Ovarian Cancer; Motolimod; Immunotherapy; PD-L1; MEDI4736; Pegylated; Liposomal; Doxorubicin; PLD; TLR-8; Durvalumab
MeSH Terms: conditions — Ovarian Neoplasms | interventions — durvalumab; liposomal doxorubicin; 1-dodecylpyridoxal; VTX-2337

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Phase 1, Dose Level 0a (Experimental): Subjects received PLD (40 mg/m^2 IV on Day 1 of every cycle) + durvalumab (3 mg/kg Q2W [equivalent to 450 mg Q4W] IV on Days 3 and 17 of every cycle) for up to 12 continuous 28-day cycles (Core Study), with extended durvalumab monotherapy permitted for subjects tolerating and benefiting from treatment. Prior to removal of motolimod from the study, subjects received motolimod (2.5 mg/m^2 SC) on Days 3, 10, and 17 of Cycles 1-3 and Days 3 and 17 of Cycles 4-12.
  Interventions: Drug: Durvalumab; Drug: Pegylated Liposomal Doxorubicin; Drug: Motolimod
- Phase 1, Dose Level 0b (Experimental): Subjects received PLD (40 mg/m^2 IV on Day 1 of every cycle) + durvalumab (1500 mg Q4W IV on Day 3 of every cycle) for up to 12 continuous 28-day cycles (Core Study), with extended durvalumab monotherapy permitted for subjects tolerating and benefiting from treatment. Prior to removal of motolimod from the study, subjects received motolimod (2.0 mg/m^2 SC) on Days 3, 10, and 17 of Cycles 1-3 and Day 3 of Cycles 4-12.
  Interventions: Drug: Durvalumab; Drug: Pegylated Liposomal Doxorubicin; Drug: Motolimod
- Phase 1, Dose Level +1 (Experimental): Subjects received PLD (40 mg/m^2 IV on Day 1 of every cycle) + durvalumab (1500 mg Q4W IV on Day 3 of every cycle) for up to 12 continuous 28-day cycles (Core Study), with extended durvalumab monotherapy permitted for subjects tolerating and benefiting from treatment. Prior to removal of motolimod from the study, subjects received motolimod (2.5 mg/m^2 SC) on Days 3, 10, and 17 of Cycles 1-3 and Day 3 of Cycles 4-12.
  Interventions: Drug: Durvalumab; Drug: Pegylated Liposomal Doxorubicin; Drug: Motolimod
- Phase 2 (Experimental): Subjects received the MTD determined in Phase 1 (Dose Level +1), comprising PLD (40 mg/m^2 IV on Day 1 of every cycle) + durvalumab (1500 mg Q4W IV on Day 3 of every cycle) for up to 12 continuous 28-day cycles (Core Study), with extended durvalumab monotherapy permitted for subjects tolerating and benefiting from treatment.
  Interventions: Drug: Durvalumab; Drug: Pegylated Liposomal Doxorubicin

INTERVENTIONS:
Drug: Durvalumab — Durvalumab is administered as an IV infusion over 60 ± 5 minutes.
  Other Names: MEDI4736
Drug: Pegylated Liposomal Doxorubicin — PLD was administered as an IV infusion in accordance with local prescribing information.
  Other Names: Doxil; Caelyx; Lipodox; PLD
Drug: Motolimod — Motolimod was administered as an SC injection. Within 30 minutes prior to each dose of motolimod, subjects were administered 650-1000 mg acetaminophen by mouth to help mitigate potential adverse events (AEs) commonly associated with the administration of motolimod (e.g., fever, myalgia). On days with concurrent motolimod and durvalumab dosing, motolimod administration occurred 30-60 minutes after the end of the durvalumab infusion. After completion of Phase 1, a protocol amendment was implemented to remove motolimod dosing from the study.
  Other Names: VTX-2337
  Arms: Phase 1, Dose Level +1; Phase 1, Dose Level 0a; Phase 1, Dose Level 0b

SUMMARY:
This is an ongoing Phase 1/2, open-label, multicenter, non-randomized study of MEDI4736 (durvalumab) in subjects with recurrent, platinum-resistant ovarian cancer who are scheduled to receive pegylated liposomal doxorubicin (PLD).The primary objective of Phase 1 is to determine the maximum tolerated dose (MTD) and safety profile, with a secondary objective to evaluate the clinical efficacy as measured by progression-free survival (PFS) rate at 6 months (PFS-6). The primary objective of Phase 2 is the evaluation of clinical efficacy as measured by PFS-6. For both phases, secondary objectives include evaluation of clinical efficacy as measured by overall response rate, PFS, and overall survival (OS), safety and tolerability, and immunological responses.

DETAILED DESCRIPTION:
In the completed Phase 1 part of the study, eligible subjects were enrolled using a standard 3 + 3 design to identify the MTD (i.e., the highest dose for which fewer than 33% of subjects experienced a dose-limiting toxicity [DLT]) of combination study treatment. All dose levels in Phase 1 included intravenous (IV) PLD (40 mg/m^2) in combination with subcutaneous (SC) motolimod (2.0 or 2.5 mg/m^2), using a starting dose of 3 mg/kg of IV durvalumab given every 2 weeks (Q2W) or 1500 mg of IV durvalumab given every 4 weeks (Q4W). All subjects in a cohort had their safety data reviewed for DLTs before proceeding with cohort expansion.

After completion of Phase 1 and determination of the durvalumab MTD to be carried forward into Phase 2, availability of data from another study (NCT01666444) indicated a lack of additive efficacy when motolimod was administered with PLD compared with PLD alone. As such, motolimod dosing was discontinued for all subjects in Study LUD2014-001 after completion of Phase 1. Subjects who had initiated treatment may have continued to receive PLD and durvalumab at their respective dose levels but must have discontinued motolimod. Thus, in the fully-accrued but ongoing Phase 2 portion of the study, subjects received only PLD (40 mg/m^2) in combination with durvalumab at the MTD determined in Phase 1 (1500 mg every 4 weeks [Q4W]).

Subjects are treated in the Core Study for an initial 12 cycles (28 days each) according to their treatment assignment. Durvalumab treatment may be extended for subjects who complete the Core Study with stable disease or better and upon agreement among the subject, Sponsor, and Investigator; extended durvalumab monotherapy may continue until confirmed disease progression, unacceptable toxicity, withdrawal of consent, or other discontinuation criteria are met.

Subjects are followed on study for 90 days after the last drug administration and off study every 3 months for 3 years from the date of the first dose of study treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must have had recurrent or persistent platinum-resistant epithelial ovarian, fallopian tube, or primary peritoneal carcinoma with measurable disease (as defined by the Response Evaluation Criteria in Solid Tumors [RECIST] 1.1.) after first or second line platinum-based chemotherapy, for which treatment with PLD was indicated. Platinum-based therapy was defined as treatment with carboplatin, cisplatin or another organoplatinum compound. Platinum-resistant was defined as having a platinum-free interval of < 12 months after first- or second-line platinum-based chemotherapy, or having disease progression while receiving second-line platinum-based chemotherapy.

   Subjects were allowed to have received, but were not required to have received:
   * one additional cytotoxic regimen and/or poly adenosine diphosphate-ribose polymerase inhibitor for management of recurrent or persistent disease.
   * biologic therapy (e.g., bevacizumab) as part of their primary treatment regimen or part of their treatment for management of recurrent or persistent disease.
2. Histologic documentation of the original primary tumor.
3. Documented radiographic disease progression < 12 months after the last dose of first- or second-line platinum-based chemotherapy.
4. Subjects in Phase 2 must have had disease amenable to biopsy and must have been willing to undergo pre- and post-treatment tumor biopsies. Optional for Phase 1.

   Note: archival tissue was requested for all subjects preferably from primary tumor site prior to cancer treatment; however, archival tissue was not a requirement for study entry.
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
6. Laboratory parameters for vital functions should have been in the normal range. Laboratory abnormalities that were not clinically significant were generally permitted, except for the following laboratory parameters, which must have been within the ranges specified, regardless of clinical significance:

   * Hemoglobin: ≥ 9 g/dL
   * Neutrophil count: ≥ 1.5 x 10^9/L
   * Platelet count: ≥ 100,000/mm^3
   * Serum creatinine: ≤ 1.5 x institutional upper limit of normal (ULN), or creatinine clearance ≥ 50 mL/min (by Cockcroft-Gault formula)
   * Serum bilirubin: ≤ 1.2 mg/dL
   * Aspartate aminotransferase (AST)/alanine aminotransferase (ALT): ≤ 2.5 x ULN
   * Alkaline phosphatase: ≤ 2.5 x ULN
7. Age ≥18 years.
8. Able and willing to give valid written informed consent.
9. Body weight > 30 kg.

Exclusion Criteria:

1. Prior exposure to doxorubicin, PLD or any other anthracycline, motolimod and other toll-like receptor agonists, durvalumab or checkpoint inhibitors, such as anti-cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) and anti-programmed cell death-1 (PD-1)/anti-programmed cell death ligand-1 (PD-L1) antibodies.
2. Subjects with platinum-refractory disease, defined as disease progression while receiving first line platinum-based therapy.
3. Clinically significant persistent immune-related adverse events following prior therapy.
4. Subjects with history or evidence upon physical examination of central nervous system disease, including primary brain tumor, seizures not controlled with standard medical therapy, any brain metastases, or, within 6 months prior to Day 1 of this study, history of cerebrovascular accident (stroke), transient ischemic attack or subarachnoid hemorrhage.
5. Subjects with clinically significant cardiovascular disease. This included:

   1. Resistant hypertension.
   2. Myocardial infarction or unstable angina within 6 months prior to Day 1 of the study.
   3. History of serious ventricular arrhythmia (i.e., ventricular tachycardia or ventricular fibrillation) or cardiac arrhythmias requiring anti-arrhythmic medications, except for atrial fibrillation that is well controlled with anti-arrhythmic medication.
   4. Baseline ejection fraction ≤ 50% as assessed by echocardiogram or multiple-gated acquisition.
   5. New York Heart Association Class II or higher congestive heart failure.
   6. Grade 2 or higher peripheral ischemia, except for brief (< 24 hours) episodes of ischemia managed non-surgically and without permanent deficit.
6. History of pneumonitis or interstitial lung disease.
7. Active, suspected or prior documented autoimmune disease (including inflammatory bowel disease, celiac disease, Wegner's granulomatosis, active Hashimoto's thyroiditis, rheumatoid arthritis, lupus, scleroderma and its variants, multiple sclerosis, myasthenia gravis). Vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger were permitted.
8. Other malignancy within 2 years prior to Day 1 of the study, except for those treated with surgical intervention only.
9. Subjects with clinical symptoms or signs of gastrointestinal obstruction and/or who required drainage gastrostomy tube and/or parenteral hydration or nutrition.
10. Known immunodeficiency or human immunodeficiency virus, Hepatitis B or Hepatitis C positivity.
11. History of severe allergic reactions to any unknown allergens or components of the study drugs.
12. Other serious illnesses (e.g., serious infections requiring antibiotics, bleeding disorders).
13. Prior treatment in any other interventional clinical trial within 4 weeks prior to Day 1 of the study.
14. Mental impairment that may have compromised compliance with the requirements of the study.
15. Lack of availability for immunological and clinical follow-up assessment.
16. Women of childbearing potential who were found to be pregnant as evidenced by positive serum pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin) or nursing. NOTE: Pregnancy tests were not required for subjects who were not of childbearing potential as defined in #17.
17. Female subjects of childbearing potential who were sexually active with a nonsterilized male partner must have used at least one highly effective method of contraception from screening, and must have agreed to continue using such precautions for 90 days after the final dose of investigational product (durvalumab). Male partners of a female subject must have used male condom plus spermicide throughout this period (from screening and for 90 days after subject's receipt of the final dose of investigational product). Cessation of birth control after this point should have been discussed with a responsible physician. Not engaging in sexual activity for the total duration of the trial and the drug washout period was an acceptable practice; however, periodic abstinence, the rhythm method, and the withdrawal method were not acceptable methods of birth control.

    Female subjects should have refrained from breastfeeding throughout the period described above.

    NOTE: For the standard of care, PLD (Doxil®, Caelyx®), the package insert advises females of reproductive potential to use effective contraception during and for 6 months after last treatment with the drug. Therefore, all subjects of childbearing potential on this study should have continued contraception use for 6 months after the last PLD administration.

    Females of childbearing potential were defined as those who were not surgically sterile (i.e., bilateral tubal ligation, bilateral oophorectomy, or complete hysterectomy) or post-menopausal.

    Females were considered post-menopausal if they had been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements applied:
    * Females < 50 years of age were considered post-menopausal if they had been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they had luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy or hysterectomy).
    * Females ≥ 50 years of age were considered post-menopausal if they had been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses > 1 year ago, had chemotherapy-induced menopause with last menses > 1 year ago, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy).

    A highly effective method of contraception was defined as one that results in a low failure rate (i.e., less than 1% per year) when used consistently and correctly. Note that some contraception methods were not considered highly effective (e.g., male or female condom with or without spermicide; female cap, diaphragm, or sponge with or without spermicide; non-copper containing intrauterine device; progestogen-only oral hormonal contraceptive pills where inhibition of ovulation is not the primary mode of action [excluding Cerazette/desogestrel which is considered highly effective]; and triphasic combined oral contraceptive pills).
18. Any condition that, in the clinical judgment of the treating physician, was likely to prevent the subject from complying with any aspect of the protocol or that may have put the subject at unacceptable risk.
19. Subjects must not have donated blood while on study and for at least 90 days following the last durvalumab treatment.
20. History of allogeneic organ transplant.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2015-12-02 (Actual); Primary Completion 2018-12-11 (Actual); Study Completion 2021-06-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George Coukos, MD, PhD, Study Chair — University of Lausanne Hospitals; Bradley J Monk, MD, Study Chair — Arizona Oncology
Locations (5):
- United States (4):
  - Research Facitlity, Phoenix, Arizona
  - Research Facility, New York, New York
  - Research Facility, Hilliard, Ohio
  - Research Facility, Providence, Rhode Island
- Research Facility, Lausanne, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R, Dancey J, Arbuck S, Gwyther S, Mooney M, Rubinstein L, Shankar L, Dodd L, Kaplan R, Lacombe D, Verweij J. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer. 2009 Jan;45(2):228-47. doi: 10.1016/j.ejca.2008.10.026. PMID 19097774
- [Background] Bohnsack O, Hoos A, Ludajic K. Adaptation of the immune related response criteria: irRECIST. Ann Oncol. 2014 Sep;25(suppl 4):iv361-iv72 [Abstract 4958]. doi: 10.1093/annonc/mdu342.23.

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 1, Dose Level 0a: Subjects received pegylated liposomal doxorubicin (PLD) (40 mg/m^2 intravenously [IV] on Day 1 of every cycle) + durvalumab (3 mg/kg every 2 weeks [Q2W, equivalent to 450 mg every 4 weeks (Q4W)] IV on Days 3 and 17 of every cycle) for up to 12 continuous 28-day cycles (Core Study), with extended durvalumab monotherapy permitted for subjects tolerating and benefiting from treatment. Prior to removal of motolimod from the study, subjects received motolimod (2.5 mg/m^2 subcutaneous [SC]) on Days 3, 10, and 17 of Cycles 1-3 and Days 3 and 17 of Cycles 4-12.
- Phase 2: Subjects received the maximum tolerated dose (MTD) determined in Phase 1, comprising PLD (40 mg/m^2 IV on Day 1 of every cycle) + durvalumab (1500 mg Q4W IV on Day 3 of every cycle) for up to 12 continuous 28-day cycles (Core Study), with extended durvalumab monotherapy permitted for subjects tolerating and benefiting from treatment.
Period: Overall Study
Arm/Group | Phase 1, Dose Level 0a | Phase 1, Dose Level 0b | Phase 1, Dose Level +1 | Phase 2
Started | 3 | 4 | 6 | 40
Completed (Completed 12 cycles of study treatment) | 1 | 1 | 2 | 9
Not Completed | 2 | 3 | 4 | 31
Not completed — Adverse Event | 0 | 1 | 0 | 4
Not completed — Progressive disease | 2 | 1 | 4 | 22
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 4
Not completed — Physician Decision | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The population comprises all subjects who received at least one dose of study treatment.
Groups:
- Phase 2: Subjects received the MTD determined in Phase 1, comprising PLD (40 mg/m^2 IV on Day 1 of every cycle) + durvalumab (1500 mg Q4W IV on Day 3 of every cycle) for up to 12 continuous 28-day cycles (Core Study), with extended durvalumab monotherapy permitted for subjects tolerating and benefiting from treatment.
- Total: Total of all reporting groups
Arm/Group | Phase 1, Dose Level 0a | Phase 1, Dose Level 0b | Phase 1, Dose Level +1 | Phase 2 | Total
Number analyzed (Participants) | 3 | 4 | 6 | 40 | 53
Age, Continuous [Median (Full Range); unit: years] | 60.0 [49 to 65] | 55.0 [33 to 63] | 62.5 [46 to 73] | 65.0 [32 to 83] | 64.0 [32 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 6 | 40 | 53
  Male | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 5 | 5
  Not Hispanic or Latino | 3 | 4 | 6 | 33 | 46
  Unknown or Not Reported | 0 | 0 | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 1 | 2
  White | 3 | 3 | 4 | 35 | 45
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 4 | 4
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 4 | 27 | 37
  Switzerland | 0 | 1 | 2 | 13 | 16
Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) at Baseline [Count of Participants; unit: Participants] — PS 0 = Fully active, able to carry on all pre-disease performance without restriction; PS 1 = Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work; PS 2 = Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours; PS 3 = Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours; PS 4 = Completely disabled; cannot carry on any selfcare; totally confined to bed or chair; PS 5 = Dead
  Participants
    0 | 3 | 2 | 5 | 34 | 44
    1 | 0 | 2 | 1 | 6 | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Treatment-emergent Adverse Events (TEAEs)
Description: The primary endpoint in Phase 1 and a secondary endpoint in Phase 2 is the safety/tolerability of study treatment. Toxicity is graded in accordance with the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 4.03. Adverse events (AEs) are reported based on clinical laboratory tests, vital signs, physical examinations, and any other medically indicated assessments, including subject interviews, from the time informed consent is signed through 90 days after the last dose of study treatment. Treatment-emergent AEs are those that occurred or worsened after administration of the first dose of study treatment.
Time Frame: Up to 3.05 years
Population: The population comprises all subjects who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1, Dose Level 0a | Phase 1, Dose Level 0b | Phase 1, Dose Level +1 | Phase 2
Number analyzed (Participants) | 3 | 4 | 6 | 40
Participants
  Any TEAE | 3 | 4 | 6 | 40
  TEAE related to any study treatment | 3 | 4 | 6 | 38
  TEAE related to durvalumab | 2 | 4 | 5 | 32
  TEAE related to PLD | 3 | 4 | 5 | 37
  TEAE related to motolimod | 3 | 4 | 6 | 1
  Serious TEAE | 0 | 2 | 1 | 23

2. Primary Outcome: Progression-free Survival Rate at 6 Months (PFS-6) by the Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as Estimated Using the Kaplan-Meier Method
Description: PFS-6 according to RECIST 1.1 is the primary endpoint in Phase 2 and a secondary endpoint in Phase 1, where PFS is measured from the date of the first dose of study treatment to the date of earliest disease progression or to the date of death, if disease progression does not occur. Per RECIST 1.1, progressive disease (PD) is defined as a ≥ 20% increase in the sum of the longest diameter of target lesions (Eisenhauer et al 2009).
Time Frame: Up to 6 months for each subject
Population: The population comprises all subjects who received at least one dose of study treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 1, Dose Level 0a | Phase 1, Dose Level 0b | Phase 1, Dose Level +1 | Phase 2
Number analyzed (Participants) | 3 | 4 | 6 | 40
percentage of participants | 33.3 [0.9 to 77.4] | 50.0 [5.8 to 84.5] | 33.3 [4.6 to 67.6] | 42.9 [27.0 to 57.8]

3. Secondary Outcome: Number of Subjects With Best Overall Tumor Response by RECIST 1.1
Description: Tumor responses were evaluated using appropriate imaging and categorized according to RECIST 1.1 at Screening (up to 14 days before the first dose of study treatment), every 3 cycles during study treatment, and during on-study follow-up approximately 3 months after the last disease assessment. Per RECIST 1.1, target lesions are categorized as follows: complete response (CR): disappearance of all target lesions; partial response (PR): ≥ 30% decrease in the sum of the longest diameter of target lesions; PD: ≥ 20% increase in the sum of the longest diameter of target lesions; stable disease (SD): small changes that do not meet above criteria (Eisenhauer et al 2009).
Time Frame: Up to 36.6 months
Population: The population comprises all subjects who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1, Dose Level 0a | Phase 1, Dose Level 0b | Phase 1, Dose Level +1 | Phase 2
Number analyzed (Participants) | 3 | 4 | 6 | 40
Participants
  CR | 0 | 0 | 0 | 4
  PR | 1 | 1 | 2 | 5
  SD | 1 | 1 | 1 | 15
  PD | 1 | 2 | 3 | 16

4. Secondary Outcome: Median PFS by RECIST 1.1 as Estimated Using the Kaplan-Meier Method
Description: PFS is measured from the date of the first dose of study treatment to the date of earliest disease progression according to RECIST 1.1 or to the date of death, if disease progression does not occur. Per RECIST 1.1, PD is defined as a ≥ 20% increase in the sum of the longest diameter of target lesions (Eisenhauer et al 2009).
Time Frame: Up to 36.6 months
Population: The population comprises all subjects who received at least one dose of study treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 1, Dose Level 0a | Phase 1, Dose Level 0b | Phase 1, Dose Level +1 | Phase 2
Number analyzed (Participants) | 3 | 4 | 6 | 40
months | 5.6 [2.7 to NA] — Upper level of confidence interval could not be estimated due to small number of patients who progressed | 5.7 [1.5 to 16.1] | 4.3 [1.2 to 16.8] | 5.5 [2.8 to 8.3]

5. Secondary Outcome: PFS-12 by RECIST 1.1 as Estimated Using the Kaplan-Meier Method
Description: as for outcome 4
Time Frame: Up to 12 months for each subject
Population: The population comprises all subjects who received at least one dose of study treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 1, Dose Level 0a | Phase 1, Dose Level 0b | Phase 1, Dose Level +1 | Phase 2
Number analyzed (Participants) | 3 | 4 | 6 | 40
percentage of participants | 33.3 [0.9 to 77.4] | 25.0 [0.9 to 66.5] | 16.7 [0.8 to 51.7] | 29.5 [15.2 to 45.2]

6. Secondary Outcome: Number of Subjects With Best Overall Tumor Response by the Immune-related Response Evaluation Criteria in Solid Tumors (irRECIST)
Description: Tumor responses were evaluated using appropriate imaging and categorized according to irRECIST at Screening (up to 14 days before the first dose of study treatment), every 3 cycles during study treatment, and during on-study follow-up approximately 3 months after the last disease assessment. Per irRECIST, measurable lesions are categorized as follows: irCR: Complete disappearance of all target lesions; irPR: ≥ 30% decrease from baseline in the total measurable tumor burden (TMTB); irPD: ≥ 20% increase from nadir in TMTB; irSD: not meeting above criteria (Bohnsack et al 2014).
Time Frame: Up to 36.6 months
Population: The population comprises all subjects who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1, Dose Level 0a | Phase 1, Dose Level 0b | Phase 1, Dose Level +1 | Phase 2
Number analyzed (Participants) | 3 | 4 | 6 | 40
Participants
  irCR | 0 | 0 | 0 | 4
  irPR | 1 | 1 | 2 | 6
  irSD | 1 | 1 | 1 | 16
  irPD | 1 | 2 | 3 | 14

7. Secondary Outcome: PFS-6 by irRECIST as Estimated Using the Kaplan-Meier Method
Description: PFS is measured from the date of the first dose of study treatment to the date of earliest disease progression according to irRECIST or to the date of death, if disease progression does not occur. Per irRECIST, irPD is defined as a ≥ 20% increase from nadir in the TMTB (Bohnsack et al 2014).
Time Frame: Up to 6 months for each subject
Population: The population comprises all subjects who received at least one dose of study treatment.
Measure: Number (95% Confidence Interval); unit: percent of participants
Arm/Group | Phase 1, Dose Level 0a | Phase 1, Dose Level 0b | Phase 1, Dose Level +1 | Phase 2
Number analyzed (Participants) | 3 | 4 | 6 | 40
percent of participants | 33.3 [0.9 to 77.4] | 50.0 [5.8 to 84.5] | 33.3 [4.6 to 67.6] | 42.6 [26.7 to 57.5]

8. Secondary Outcome: PFS-12 by irRECIST as Estimated Using the Kaplan-Meier Method
Description: as for outcome 7
Time Frame: Up to 12 months for each subject
Population: The population comprises all subjects who received at least one dose of study treatment.
Measure: Number (95% Confidence Interval); unit: percent of participants
Arm/Group | Phase 1, Dose Level 0a | Phase 1, Dose Level 0b | Phase 1, Dose Level +1 | Phase 2
Number analyzed (Participants) | 3 | 4 | 6 | 40
percent of participants | 33.3 [0.9 to 77.4] | 25.0 [0.9 to 66.5] | 16.7 [0.8 to 51.7] | 33.4 [18.8 to 48.7]

9. Secondary Outcome: Median PFS by irRECIST as Estimated Using the Kaplan-Meier Method
Description: as for outcome 7
Time Frame: Up to 36.6 months
Population: The population comprises all subjects who received at least one dose of study treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 1, Dose Level 0a | Phase 1, Dose Level 0b | Phase 1, Dose Level +1 | Phase 2
Number analyzed (Participants) | 3 | 4 | 6 | 40
months | 5.6 [2.7 to NA] — Upper limit of confidence interval was not estimable due to small number of patients with events. | 5.7 [1.5 to 16.1] | 4.3 [1.2 to 16.8] | 5.5 [3.0 to 8.3]

10. Secondary Outcome: Median Overall Survival (OS) as Estimated Using the Kaplan-Meier Method
Description: After completion of treatment, all subjects are followed for survival every 3 months for up to 3 years following initiation of study treatment or or for subjects continuing treatment, completion of study treatment whichever was longer. OS is measured from the date of the first dose of study treatment to the date of death or last follow-up. Subjects lost to follow-up are censored on the date when they were last known to be alive.
Time Frame: Up to 36.6 months
Population: The population comprises all subjects who received at least one dose of study treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 1, Dose Level 0a | Phase 1, Dose Level 0b | Phase 1, Dose Level +1 | Phase 2
Number analyzed (Participants) | 3 | 4 | 6 | 40
months | 27.7 [11.8 to NA] — Upper limit of confidence interval was not estimable due to small number of patients with events. | NA [4.2 to NA] — Median OS for Phase 1, Dose Level 0b and upper limit of confidence interval were not estimable due to small number of patients with events. | 12.8 [4.0 to NA] — Upper limit of confidence interval was not estimable due to small number of patients with events. | 17.6 [11.6 to NA] — Upper limit of confidence interval was not estimable due to small number of patients with events.

ADVERSE EVENTS:
Time Frame: All AEs occurring between the signing of informed consent and the off-study date (i.e., through 90 days after the last dose of study treatment [up to 3.05 years]) are documented, regardless of the causal relationship to study drug. AEs that occur or worsen in severity after the first dose of study treatment are considered treatment emergent (i.e., TEAEs).
Description: AE documentation includes onset/resolution dates, severity using the NCI CTCAE (version 4.03), seriousness, relationship to study drug, study drug action taken, treatment, and outcome. In summaries, preferred terms are counted only once per subject at the maximum reported grade.
Arm/Group | Phase 1, Dose Level 0a | Phase 1, Dose Level 0b | Phase 1, Dose Level +1 | Phase 2
All-Cause Mortality (participants affected / at risk) | 2/3 | 2/4 | 4/6 | 21/40
Serious Adverse Events (participants affected / at risk) | 0/3 | 2/4 | 1/6 | 23/40
Other Adverse Events (participants affected / at risk) | 3/3 | 4/4 | 6/6 | 40/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1, Dose Level 0a (N=3) | Phase 1, Dose Level 0b (N=4) | Phase 1, Dose Level +1 (N=6) | Phase 2 (N=40)
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 3
Aphasia (Nervous system disorders) | 0 | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1
Bacterial translocation (Infections and infestations) | 0 | 0 | 0 | 1
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2
Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2
General physical health deterioration (General disorders) | 0 | 0 | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 1 | 2
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Lung infection (Infections and infestations) | 0 | 0 | 0 | 2
Lymphadenectomy (Surgical and medical procedures) | 0 | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 3
Nutritional condition abnormal (Investigations) | 0 | 0 | 0 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2
Pleural fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 3
Rectal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 2
Subileus (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 1
Urinary tract obstruction (Renal and urinary disorders) | 0 | 1 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Wound complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Radiculitis (Nervous system disorders) | 0 | 0 | 0 | 1
Tumour excision (Surgical and medical procedures) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1, Dose Level 0a (N=3) | Phase 1, Dose Level 0b (N=4) | Phase 1, Dose Level +1 (N=6) | Phase 2 (N=40)
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 2 | 9
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 8
Alanine aminotransferase increased (Investigations) | 0 | 1 | 1 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 5
Amylase increased (Investigations) | 0 | 0 | 0 | 7
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 7
Anal fissure (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Anal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 2 | 0 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 8
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 1 | 2
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 3
Blood folate decreased (Investigations) | 0 | 1 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 1 | 1
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 1
Catheter site pain (General disorders) | 0 | 0 | 0 | 2
Chest discomfort (General disorders) | 0 | 1 | 1 | 0
Chills (General disorders) | 2 | 2 | 6 | 4
Confusional state (Psychiatric disorders) | 1 | 0 | 0 | 1
Conjunctival ulcer (Eye disorders) | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 2 | 2 | 11
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 11
C-reactive protein increased (Investigations) | 0 | 0 | 1 | 5
Cystitis (Infections and infestations) | 0 | 0 | 0 | 2
Decreased appetite (Metabolism and nutrition disorders) | 0 | 3 | 1 | 9
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 1
Depression (Psychiatric disorders) | 0 | 0 | 0 | 3
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 2 | 10
Dry eye (Eye disorders) | 1 | 2 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 1 | 3
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 2 | 1 | 4
Dysgeusia (Nervous system disorders) | 0 | 0 | 1 | 3
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 2 | 3
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Dysphonia psychogenic (Nervous system disorders) | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 8
Dysuria (Renal and urinary disorders) | 0 | 0 | 1 | 1
Embolism (Vascular disorders) | 0 | 1 | 0 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 3
Eye pain (Eye disorders) | 0 | 1 | 0 | 0
Fatigue (General disorders) | 3 | 3 | 4 | 21
Feeling cold (General disorders) | 0 | 0 | 1 | 0
Folliculitis (Infections and infestations) | 1 | 1 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 1 | 1
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 2 | 5
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 1 | 1 | 0
Headache (Nervous system disorders) | 2 | 2 | 1 | 4
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 1 | 1 | 0 | 4
Hyperthyroidism (Endocrine disorders) | 2 | 0 | 1 | 4
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 6
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 7
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 5
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 3
Hypotension (Vascular disorders) | 0 | 0 | 1 | 3
Hypothyroidism (Endocrine disorders) | 1 | 2 | 2 | 3
Influenza (Infections and infestations) | 0 | 0 | 1 | 0
Influenza like illness (General disorders) | 3 | 1 | 0 | 2
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 3
Injection site discolouration (General disorders) | 0 | 0 | 1 | 0
Injection site erythema (General disorders) | 0 | 1 | 0 | 0
Injection site pain (General disorders) | 0 | 0 | 1 | 0
Injection site reaction (General disorders) | 3 | 3 | 5 | 0
Injection site vesicles (General disorders) | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 2 | 0 | 7
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Lipase increased (Investigations) | 0 | 0 | 0 | 6
Lymphocyte count decreased (Investigations) | 0 | 0 | 1 | 10
Lymphoedema (Vascular disorders) | 1 | 0 | 0 | 1
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Mucosal infection (Infections and infestations) | 0 | 0 | 1 | 4
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 5
Nausea (Gastrointestinal disorders) | 1 | 4 | 3 | 19
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 2
Neutrophil count decreased (Investigations) | 0 | 1 | 1 | 2
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 3
Oedema peripheral (General disorders) | 0 | 0 | 0 | 2
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 2
Oral pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2
Otitis media (Infections and infestations) | 0 | 1 | 0 | 1
Pain (General disorders) | 0 | 0 | 0 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 2 | 1 | 3 | 23
Palpitations (Cardiac disorders) | 0 | 1 | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 1 | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1 | 0 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2
Platelet count decreased (Investigations) | 0 | 0 | 0 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 3
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 1 | 1
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 5
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 11
Pyelonephritis (Infections and infestations) | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 2 | 2 | 5 | 10
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 6
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 | 2 | 2 | 19
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Renal colic (Renal and urinary disorders) | 0 | 0 | 1 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 0 | 3
Respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 2
Sensation of foreign body (General disorders) | 0 | 1 | 1 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 2
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 1 | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 1 | 3 | 2
Skin induration (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 3
Stomatitis (Gastrointestinal disorders) | 2 | 2 | 4 | 18
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 0 | 2
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 2
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 3
Urinary tract pain (Renal and urinary disorders) | 1 | 0 | 0 | 2
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Vaginal discharge (Reproductive system and breast disorders) | 0 | 1 | 0 | 1
Viral skin infection (Infections and infestations) | 0 | 1 | 0 | 0
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2
Vomiting (Gastrointestinal disorders) | 0 | 3 | 3 | 11
Vulvovaginal candidiasis (Infections and infestations) | 0 | 0 | 1 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 6
Weight increased (Investigations) | 1 | 0 | 1 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 1 | 3
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Catheter site rash (General disorders) | 0 | 0 | 1 | 0
Malaise (General disorders) | 0 | 0 | 0 | 2
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 2
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2017-09-08): https://cdn.clinicaltrials.gov/large-docs/59/NCT02431559/Prot_000.pdf
  • Statistical Analysis Plan (2019-01-08): https://cdn.clinicaltrials.gov/large-docs/59/NCT02431559/SAP_001.pdf